CLINICAL TRIAL: NCT01187251
Title: Incidence of Tinnitus Amongst Teenagers and Young Adults mp3 Users
Status: Completed | Type: Observational
Sponsor: Faculdade de Medicina de Valenca (Other)
Other Study IDs: tinnitus and mp3 players
Record Dates: First submitted 2010-08-23; First posted 2010-08-24 (Estimated); Last update posted 2010-08-24 (Estimated); Status verified 2010-02

CONDITIONS: Tinnitus
Keywords: tinnitus; mp3 players; noise induced hearing loss; high frequencies audiometry; acoustic otoemissions
MeSH Terms: conditions — Tinnitus; Hearing Loss, Noise-Induced

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1 - mp3 users: Subjects who have been using mp3 players for at least 1 hour per day for at least 1 year
- Group 2 - mp3 non-users: Subjects who does not listen regularly to mp3 music

SUMMARY:
The aim of this study is to compare the incidence of tinnitus between mp3 users and non-users, aged between 15 and 30 years old. 100 patients will be recruited in Valença secondary schools. High frequency audiometry and otoacoustic emissions will be performed.Tinnitus patients will complete the Tinnitus Handicap Inventory questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* 15 to 30 years old
* A-n tympanogram

Exclusion Criteria:

* muscular tinnitus
* vascular tinnitus
* somatosensorial tinnitus
* concomitant TMJ disorders
* external and middle ear diseases
* professional or recreative exposure to other noise sources other than mp3 players

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: teenagers and young adults (15 to 30 years old)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2009-08; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - caculdade de Medicina de Valença, Valença, Rio de Janeiro
  - OTOSUL,Otorrinolaringologia Sul-Fluminense, Volta Redonda, Rio de Janeiro